CLINICAL TRIAL: NCT04110223
Title: Validation Studies of Biomarkers for Precision Radiation Oncology in Locally Advanced Solid Tumors
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shandong Cancer Hospital and Institute (Other)
Responsible Party: Principal Investigator, Jinming Yu, President, Shandong Cancer Hospital and Institute
Other Study IDs: GBRT-043
Record Dates: First submitted 2019-06-12; First posted 2019-10-01 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Radiation Toxicity; Advanced Cancer; Radiosensitivity
Keywords: radiotherapy; radiosensitivity; radiation toxity; NGS
MeSH Terms: conditions — Radiation Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — tumor biopsy samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- non-smell cell lung cancer (NSCLC): Advanced NSCLC patients receiving radiotherapy or chemo-radiotherapy
  Interventions: Genetic: next generation sequence
- Rectal cancer: Rectal cancer patients receiving neoadjuvant radiotherapy or chemo-radiotherapy
  Interventions: Genetic: next generation sequence
- Smell cell lung cancer (SCLC): SCLC patients receiving radiotherapy or chemo-radiotherapy
  Interventions: Genetic: next generation sequence
- Esophageal cancer: Esophageal cancer patients receiving radiotherapy or chemo-radiotherapy
  Interventions: Genetic: next generation sequence
- Cervical cancer: Cervical cancer patients receiving radiotherapy or chemo-radiotherapy
  Interventions: Genetic: next generation sequence
- Liver cancer: Liver cancer atients receiving radiotherapy or chemo-radiotherapy
  Interventions: Genetic: next generation sequence

INTERVENTIONS:
Genetic: next generation sequence — targeted NGS of patients' pretreatment tumor biopsy samples using a 474-gene panel, which covers cancer- and radio-sensitivity-related mutations and SNPs.

SUMMARY:
Despite the common application of radiotherapy in cancer treatment, the prediction of radiosensitivity and treatment response has not yet entered the era of precision medicine. Therefore, development of genome-based methods for predicting radiosensitivity and treatment response is a central goal of radiation oncology. In the previous study, the investigators have identified a set of novel potential biomarkers associated with radiosensitivity and recurrence，through correlating patients' genomic profiles with toxicity, disease progression and overall survival after RT.

DETAILED DESCRIPTION:
Researchers have long recognized that individual differences in sensitivity to radiation are caused by genetic variations and implicated multiple key pathways that might explain radiation toxicity. Normal tissue toxicity is a complex trait that involves the combined effect of a multitude of genes and pathways, and also dynamic interactions with the evolving cancer genome. The effect size of any individual factor is likely small. As a consequence, candidate gene approach and genome-wide association studies rarely lead to the identification of genetic determinants of radiation toxicity. Targeted next-generation sequencing (NGS), on the other hand, has become increasingly routine in the clinic and would allow simultaneous assessment of multiple genetic alterations.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with locally advanced solid tumors (lung cancer, esophageal cancer, rectal cancer (neoadjuvant), cervical cancer, nasopharyngeal carcinoma cancer and liver cancer) identified by cytology and pathology;
2. Patients need conventional fractionation and adequate radiotherapy;
3. Age ≥ 18 years old, male and female;
4. Expected survival time ≥ 12 weeks;
5. PS score 0-2 within 2 weeks before admission to the group;
6. There are tumor tissue samples and blood samples can be used for NGS inspection;
7. Patients volunteered to join this study, sign informed consent, provide all diagnosis and treatment data after cancer diagnosis before entering the group, good compliance, cooperate with follow-up.

Exclusion Criteria:

1. The patient's previous radiation therapy leads to overlapping potential fields;
2. Stage IV patients and stage I patients to be treated with SBRT
3. The patient cannot receive regular imaging examinations;
4. Any serious or uncontrolled signs of systemic disease that the investigator believes may significantly affect the patient's risk/benefit balance, including hepatitis B, hepatitis C, and human immunodeficiency virus;
5. The researcher believes that it is not suitable for the group.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in the study with locally advanced solid tumors undergoing conventional fractionation or preoperative neoadjuvant radiotherapy (except stage IV patients and stage I patients to be treated with SBRT), including lung cancer, esophageal cancer, rectal cancer (neoadjuvant), cervical cancer, nasopharyngeal carcinoma and liver cancer
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2018-10-08 (Actual); Primary Completion 2021-10-08 (Estimated); Study Completion 2021-10-08 (Estimated)

PRIMARY OUTCOMES:
TTP | 2 years
  Time to progression
OS | 2 years
  Time to death

CONTACTS AND LOCATIONS:
Overall Officials: Jinming Yu, Ph.D, Principal Investigator — Shandong Cancer Hospital and Institute
Locations (1):
- Shandong Cancer Hospital and Institute, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No